CLINICAL TRIAL: NCT01635699
Title: Effect of Modified Fujita Technique Uvulopalatoplasty on Oxidative DNA Damage Levels in Patients With Obstructive Sleep Apnea SyndromE
Brief Title: Effect of Modified Fujita Technique Uvulopalatoplasty on Oxidative DNA Damage Levels in Patients With Obstructive Sleep Apnea SyndromE (OSAS)
Status: Completed | Type: Observational
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Vural Fidan, operating surgeon doctor, Erzurum Regional Training & Research Hospital
Other Study IDs: ATUNI-1
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: DNA oxidation; obstructive sleep apnea; lipid peroxidation; oxidative stresses
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the possible effects of uvulopalatopharngoplasty (UPPP) -which is a a therapy used on patients with Obstructive sleep apnea syndrome (OSAS- on oxidative damage.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a sydrome which has characteristic upper way obstruction and a decrease in blood oxygen saturation as sleeping. uvulopalatopharngoplasty (UPPP)is one of the surgical approaches applied to the patients with OSAS, since the oxidative damage markers have been found high in patients with OSAS. Although antioxidant levels were higher in patients with OSAS than those in normal population, there is report about the effect of UPPP on antioxidant status in patients with OSAS. We performed this study to confirm whether is there a We performed the present study to confirm whether there is a relationship between the OSAS and oxidative damage before and after UPPP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent uvulopalatopharngoplasty (UPPP)for Obstructive sleep apnea syndrome (OSAS)

Exclusion Criteria:

* Anormal nasopharyngeal computed tomography, chronic diseases such as diabetes mellitus, hypertension etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent uvulopalatopharngoplasty (UPPP)for Obstructive sleep apnea syndrome (OSAS) at the otolaryngology department of our hospital in Erzurum, Turkey.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: vural fidan, operating surgeon doctor, Principal Investigator — eskisehir yunus emre state hospital (still works here)
Locations (1):
- Erzurum Regional Educational Researh Hospital, Erzurum, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Bakan E, Fidan V, Alp HH, Baygutalp NK, Cokluk E. Effect of Modified Fujita Technique Uvulopalatoplasty on Oxidative DNA Damage Levels in Patients With Obstructive Sleep Apnea Syndrome. J Craniofac Surg. 2015 Jul;26(5):e392-6. doi: 10.1097/SCS.0000000000001870. PMID 26163849